CLINICAL TRIAL: NCT00167661
Title: Campath-1H Induction to Allow Steroid Free Immunosuppression in Pediatric Renal Transplantation
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Enrollment suspended pending protocol revision to change study to observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0661; H-2003-0493 (Other: UW IRB); A536758 (Other: UW Madison); SMPH/PEDIATRICS/PEDIATRICS (Other: UW Madison)
Record Dates: First submitted 2005-09-11; First posted 2005-09-14 (Estimated); Results first posted 2020-09-21 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-08

CONDITIONS: Disorder Related to Renal Transplantation
Keywords: living or deceased donor renal transplant recipient
MeSH Terms: interventions — Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Campath 1-H (Experimental): Campath 1-H
  Interventions: Drug: Campath-1H

INTERVENTIONS:
Drug: Campath-1H — two intravenous 20mg/m2/doses, the first on the day of transplant and the second dose on day 1 post transplant
  Other Names: Alemtuzumab

SUMMARY:
The purpose of this study is to determine whether Campath-1H induction and the associated lymphocyte depletion will permit long-term rejection-free renal allograft survival in the absence of ongoing corticosteroid administration.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be a single-organ recipient (kidney only)
* Participants who are receiving their first living donor or deceased donor transplant

Exclusion Criteria:

* Participants who are recipients of HLA-identical living-donor renal transplants
* Participants with a PRA value > 10% within 30 days prior to the transplant
* Participants who have received a multi-organ transplant
* Participants who are who are positive for hepatitis C, hepatitis B surface antigen or HIV
* Participants who have received an investigational drug within 6 weeks of study entry
* Participants who have a previous history of, or who currently have, malignancies and/or lymphoma
* Participants who have received corticosteroids within three months of transplantation
* Participants who are 3rd transplant recipients
* Female participants who are pregnant or lactating. Fertile female participants who are sexually active must agree to use an acceptable method of birth control during the study

Ages: 18 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2004-06; Primary Completion 2011-12 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon M Bartosh, MD, Study Chair — University of Wisconsin, Madison; Sharon M Bartosh, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Campath 1-H
Started | 33
Completed | 33
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Campath 1-H
Number analyzed (Participants) | 33
Age, Continuous [Mean (Full Range); unit: years] | 11.8 [2.1 to 18.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 32
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 26
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Graft Rejection
Time Frame: at 1, 3, 6, 12, and 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Campath 1-H
Number analyzed (Participants) | 33
Participants
  1 month | 0
  3 months | 2
  6 months | 6
  12 months | 10
  24 months | 11

2. Primary Outcome: Participant Graft Survival
Time Frame: at 6, 12, and 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Campath 1-H
Number analyzed (Participants) | 33
Participants
  6 months | 32
  12 months | 32
  24 months | 32

3. Secondary Outcome: Estimated Glomerular Filtration Rate (EGFR)
Description: Measure of renal function
Time Frame: at 1, 6, 12 and 24 months
Population: One participant was on dialysis at 2 years, not included in the analysis
Measure: Mean (Full Range); unit: ml/min/1.73m^2
Arm/Group | Campath 1-H
Number analyzed (Participants) | 33
ml/min/1.73m^2
  1 month | 91.5 [37 to 150]
  6 months | 88.4 [15 to 161]
  12 months | 85.8 [11 to 139]
  24 months: number analyzed (Participants) | 32
  24 months | 77.4 [25 to 126]

4. Secondary Outcome: Number of Participants With Infection
Description: Cytomegalovirus(CMV), Epstein Barr Virus (EBV) BK Virus (BK)
Time Frame: up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Campath 1-H
Number analyzed (Participants) | 33
Participants
  BK Nephropathy | 2
  BK Viremia | 10
  BK Viruria | 12
  CMV Viremia | 4
  CMV disease | 0
  EBV Viremia | 1
  EBV disease | 0

5. Secondary Outcome: Number of Participants With Malignancy
Time Frame: up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Campath 1-H
Number analyzed (Participants) | 33
Participants | 0

6. Secondary Outcome: Growth Post-transplant Reported by Height Z Score
Description: A z-score (aka, a standard score) indicates how many standard deviations an element is from the mean, in this case, height. A score of '0' is equal to the mean, a score less than 0 is less than the mean, and a score greater than 0 is greater than the mean.
Time Frame: up to 24 months
Population: One participant was on dialysis at 2 years, not included in the analysis
Measure: Mean (Full Range); unit: z-score
Arm/Group | Campath 1-H
Number analyzed (Participants) | 33
z-score
  baseline | -0.99 [-5.0 to 1.25]
  12 months | -0.41 [-3.06 to 1.40]
  24 months: number analyzed (Participants) | 32
  24 months | -0.35 [-2.31 to 1.33]

7. Secondary Outcome: Number of Participants With Hypertension
Time Frame: up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Campath 1-H
Number analyzed (Participants) | 33
Participants | 27

8. Secondary Outcome: Number of Participants With Hyperlipidemia
Time Frame: up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Campath 1-H
Number analyzed (Participants) | 33
Participants | 0

9. Secondary Outcome: Participant Survival
Time Frame: at 6, 12, and 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Campath 1-H
Number analyzed (Participants) | 33
Participants
  6 months | 33
  12 months | 33
  24 months | 33

10. Secondary Outcome: Number of Participant With Diabetes Mellitus
Time Frame: up to 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Campath 1-H
Number analyzed (Participants) | 33
Participants | 0

ADVERSE EVENTS:
Time Frame: up to 24 months
Arm/Group | Campath 1-H
All-Cause Mortality (participants affected / at risk) | 0/33
Serious Adverse Events (participants affected / at risk) | 2/33
Other Adverse Events (participants affected / at risk) | 29/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Campath 1-H (N=33)
Pyuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Increase Creatinine (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Campath 1-H (N=33)
Fever (General disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 4
Gingivitis (Infections and infestations) | 1
influenza (Infections and infestations) | 3
Diarrhea (Gastrointestinal disorders) | 7
Urinary Tract Infection (Infections and infestations) | 2
Pseudomonas bacteremia (Infections and infestations) | 1
Varicella (Infections and infestations) | 2
Dehydration (General disorders) | 3
Ureteral Stricture (Renal and urinary disorders) | 1
Pneumonia (Infections and infestations) | 3
Seizure (Nervous system disorders) | 1
Small Bowel Obstruction (Gastrointestinal disorders) | 2
Pyelonephritis (Renal and urinary disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Epigastric Pain (Gastrointestinal disorders) | 1
Hydroureter (Renal and urinary disorders) | 1
Elevated Creatinine (Renal and urinary disorders) | 9
Increased Proteinuria (Renal and urinary disorders) | 3
Pyuria (Renal and urinary disorders) | 1
Renal Insufficiency (Renal and urinary disorders) | 1
Urinary Eosinophils (Renal and urinary disorders) | 1
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 2
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 3
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 3
Tonsillar cervical, axillary, inguinal hypertrophy (Immune system disorders) | 7
Anemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hyperphosphatemia (Metabolism and nutrition disorders) | 1
Weight Loss (Metabolism and nutrition disorders) | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1
Mouth Ulcers (Skin and subcutaneous tissue disorders) | 2
Hives (Immune system disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 5
Chest Pain (General disorders) | 1
fatigue (General disorders) | 1
Nausea and Vomiting (Gastrointestinal disorders) | 3
Headache (General disorders) | 2
Joint Pain (General disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 9
Eosinophilia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 5
Lymphoid hyperplasia (Blood and lymphatic system disorders) | 1
Fine tremor at rest (Nervous system disorders) | 1
Fracture L5 (Injury, poisoning and procedural complications) | 1
High Blood Pressure (Vascular disorders) | 2
Hepatosplenomegaly (Hepatobiliary disorders) | 1
Left ventricular hypertrophy (Cardiac disorders) | 1
Ottis Media (Ear and labyrinth disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes